CLINICAL TRIAL: NCT00327457
Title: Coordinated Endoscopic Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Association of Schools of Public Health (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: S1796-21/23 (NCE)
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Preventive Health Services
Keywords: colorectal cancer screening; sigmoidoscopy; colonoscopy
MeSH Terms: interventions — Insemination, Artificial, Heterologous; Physicians' Offices

INTERVENTIONS:
Behavioral: Help with physician office and patient management
Behavioral: Tailored physician recommendation letter

SUMMARY:
The investigators aim to use a randomized design to test the effects of 1) tailored physician recommendations, relative to non-specific recommendations, and 2) coordinated physician office management systems on patient adherence to colorectal cancer screening recommendations.

DETAILED DESCRIPTION:
The investigators aim to use a randomized design to test the effects of 1) tailored physician recommendations, relative to non-specific recommendations, and 2) coordinated physician office management systems on patient adherence to colorectal cancer screening recommendations.

To accomplish these aims, the investigators propose 1) to use existing physician practice-based computerized patient registration systems to define populations of 50 to 79 year-old pri-mary care patients, 2) to use mailed questionnaires to determine colorectal cancer risk factor status and prior colorectal cancer screening history, 3) to use responses from mailed questionnaires to identify persons not adhering to colorectal cancer screening guidelines, 4) to use computer driven algorithms to help physicians prepare and deliver individually tailored and written colorectal cancer screening recommendations, and 5) to develop, implement, and evaluate a centralized service for delivering high quality screening flexible sigmoidoscopy.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* history of colorectal cancer or polyps
* flexible sigmoidoscopy within five years of enrollment
* barium enema within five years of enrollment
* colonoscopy within five years of enrollment

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2002-06; Study Completion 2005-03

PRIMARY OUTCOMES:
Medical record verified flexible sigmoidoscopy or colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Joel L. Weissfeld, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Ling BS, Schoen RE, Trauth JM, Wahed AS, Eury T, Simak DM, Solano FX, Weissfeld JL. Physicians encouraging colorectal screening: a randomized controlled trial of enhanced office and patient management on compliance with colorectal cancer screening. Arch Intern Med. 2009 Jan 12;169(1):47-55. doi: 10.1001/archinternmed.2008.519. PMID 19139323